CLINICAL TRIAL: NCT02680353
Title: The Perioperative Analgesic Efficiency of Bilateral Superficial Cervical Plexus Block in Patients With Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assist.Prof., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-KAEK-055
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Block
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Active Comparator): Patients received bilateral superficial cervical plexus block before operation
  Interventions: Procedure: Bilateral superficial cervical plexus block
- Control group (No Intervention): Patients received no intervention before operation

INTERVENTIONS:
Procedure: Bilateral superficial cervical plexus block — A kind of anesthetic nerve block type performed to block the nerve function temporarily by administrating local anesthetics through the trajectory of the nerve.
  Arms: Study group

SUMMARY:
To determine the postoperative analgesic efficiency of bilateral superficial plexus block, patients are divided into two groups. Study group received bilateral superficial plexus block, where control had none. Visual analog scale, opioid consumption and presence of nausea-vomiting are recorded.

DETAILED DESCRIPTION:
Bilateral superficial cervical plexus block has successfully been demonstrated to provide an efficient analgesia in patients with thyroidectomy, parathyroidectomy, carotis end-arterectomy. The present study is aimed to investigate the intraoperative hemodynamic responses, anesthetic and analgesic consumption, and postoperative recovery quality of bilateral superficial cervical plexus block in patients with total thyroidectomy. After approval, patients enrolled in the study is invited to complete the Pain Catastrophizing Scale questionnaire. Patients are divided into two groups by computer-based randomization technique as control and study group. After standard monitorization, anesthesia induction and tracheal intubation, bilateral superficial cervical plexus block is performed to study group and no intervention to control group. At the end of the operation all patients received paracetamol 1 gr intravenous. In postoperative period, visual analog scale values, opioid consumption, presence of nausea-vomiting, anti-emetic usage or any other complications are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Planned to undergo thyroidectomy
* An American Society of Anesthesiologists score of 1 or 2

Exclusion Criteria:

* Severe cardiovascular disease
* Psychiatric diseases
* Difficult intubation
* Rejected to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | one time in postoperative period for one year

SECONDARY OUTCOMES:
Presence of nausea-vomiting | In postoperative period for one year
Mean arterial pressure | In both intraoperative and postoperative period for one year
Heart rate | In both intraoperative and postoperative period for one year
Antiemetic usage | postoperative period for one year
respiratory rate | postoperative period for one year
opioid consumption | During postoperative period for one year

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Assist.Prof, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No